CLINICAL TRIAL: NCT06654375
Title: Thrombectomy Versus Best Medical Management in Large Vessel Occlusion Stroke Patients Presenting Beyond 24 Hours and With Presence of Collateral Flow on CT Angiography: A Multicentre, Open-label, Registry-linked, Randomised Controlled Trial
Brief Title: Thrombectomy Versus Best Medical Management in Large Vessel Occlusion Stroke Patients Presenting Beyond 24 Hours and With Presence of Collateral Flow on CT Angiography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ming Wei, Chief Physician, Tianjin Huanhu Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: tjhh202410
Record Dates: First submitted 2024-10-14; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Stroke Acute; Thrombectomy; Medical Treatment; Large Vessel Occlusion
Keywords: CTA; Endovascular Thrombectomy; Acute Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular thrombectomy (Experimental)
  Interventions: Procedure: Endovascular Thrombectomy
- Best Medical Management (No Intervention)

INTERVENTIONS:
Procedure: Endovascular Thrombectomy — Endovascular thrombectomy (EVT) in this clinical trial involves the mechanical removal of a thrombus from a blocked large cerebral artery using specialized devices like stent retrievers or aspiration catheters. Key distinguishing features of this EVT protocol include:
  * Extended Time Window: Unlike standard EVT, which is typically performed within 24 hours after symptom onset, this intervention targets patients presenting beyond 24 hours.
  * Collateral Circulation Assessment: Multi-phase CT angiography (CTA) is employed to evaluate collateral flow, prioritizing patients with favorable collateral grades. This selection process helps ensure the identification of patients most likely to benefit from EVT despite the late presentation.
  Arms: Endovascular thrombectomy

SUMMARY:
The goal of this clinical trial is to investigate if endovascular treatment (EVT) can effectively treat patients with large vessel occlusion (LVO) who present beyond the typical 24-hour window after symptom onset. The main questions it aims to answer are:

* Can EVT improve functional independence at 90 days for patients treated after 24 hours?
* What is the safety profile of EVT in this delayed treatment group compared to best medical management (BMM)? Researchers will compare EVT outcomes in patients presenting after 24 hours to those receiving BMM to see if EVT offers significant benefits.

Participants will:

* Receive either EVT or BMM based on their eligibility.
* Undergo CT angiography to assess collateral circulation and to confirm the presence of LVO.
* Be followed for 90 days to evaluate functional outcomes and safety measures.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmation of ICA or MCA-M1 occlusion, as detected by MRA or CTA, with carotid occlusions potentially occurring in either the cervical or intracranial regions, and the possibility of accompanying tandem MCA lesions.
2. Demonstration of moderate to good collateral flow, as evidenced by CTA imaging.
3. The patient must be aged 18 years or older.
4. The baseline NIHSSS score is equal to or greater than 2, and this score remains equal to or greater than 2 immediately prior to randomization.
5. Endovascular treatment can be initiated (via femoral puncture) within a window of 24 to 72 hours from the onset of the stroke. The onset of the stroke is defined as the time the patient was last known to be at their neurologic baseline (patients with wake-up strokes are eligible if they meet the aforementioned time constraints).
6. There must be no significant pre-stroke disability, as indicated by a pre-baseline modified Rankin Scale score of 0-2.
7. The patient must be willing and able to return for the protocol-required follow-up visits.
8. The patient or their legally authorized representative must have signed the Informed Consent form.

Exclusion Criteria:

1. The subject has a serious, advanced, or terminal illness (as determined by the investigator) or a life expectancy of less than six months.
2. The subject has a pre-existing medical, neurological, or psychiatric disease that would interfere with neurological or functional evaluations, or is already participating in another drug or device study.
3. The subject is pregnant.
4. The subject has contraindications for both MRI and CT contrast that prevent an MRI or CT contrast perfusion study. The hospital's local standard criteria should be applied to determine if contraindications exist.
5. The subject has a known allergy to iodine and has previously been refractory to pretreatment medications.
6. The subject has been treated with tPA more than 4.5 hours after the last known well time.
7. The subject has a known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency, or has recently undergone oral anticoagulant therapy with an INR greater than 3.
8. The subject has symptoms consistent with stroke in multiple locations.
9. The subject has seizures at stroke onset, which makes the diagnosis of stroke doubtful and precludes obtaining an accurate baseline NIHSS assessment.
10. The subject has a baseline blood glucose level of less than 50mg/dL (2.78 mmol) or greater than 400mg/dL (22.20 mmol).
11. The subject has a baseline platelet count of less than 50,000/uL.
12. The subject has severe, sustained hypertension (Systolic Blood Pressure >185 mmHg or Diastolic Blood Pressure >110 mmHg) that is not treatable with medications.
13. The subject is currently participating in another investigational drug or device study or registry.
14. The subject is presumed to have a septic embolus, suspicion of bacterial endocarditis, or cerebral vasculitis.
15. The subject has had clot retrieval attempted using a neurothrombectomy device within 24 hours of symptom onset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale | 90 days (± 14 days)
  a 7-point scale ranging from 0 (no symptoms) to 6 (death)

SECONDARY OUTCOMES:
extended treatment in cerebral ischemia (eTICI) score | during EVT procedure
recanalization rate | 24 hours after randomization, assessed using Computed Tomography Angiography (CTA) or Magnetic Resonance Angiography (MRA)
score on the NIHSS | 24 hours after randomization, 5 to 7 days after randomization, or at discharge, whichever occurs first
final infarct volume on MRI | 24 hours after randomization on MRI
dichotomized mRS score of 0-1 vs 2-6 | at 90 days
dichotomized mRS score of of 0-2 vs 3-6 | at 90 days
dichotomized mRS score of 0-3 vs 4-6 | at 90 days
death | at 90 days
Score on the Barthel Index | at 90 days
Score on the EQ-5D-5L | at 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No